CLINICAL TRIAL: NCT06589310
Title: Falcon - The Exact Sciences Multicancer Early Detection (MCED) Real World Evidence (RWE) Registry
Brief Title: Falcon Real World Evidence Registry
Status: Recruiting | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: EXAS 2022-02
Record Dates: First submitted 2024-08-19; First posted 2024-09-19 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Multicancer Early Detection (MCED) cohort
  Interventions: Device: Exact Sciences Multicancer Early Detection (MCED) Test

INTERVENTIONS:
Device: Exact Sciences Multicancer Early Detection (MCED) Test — Exact Sciences MCED test, is a qualitative in vitro diagnostic (IVD) for the detection of alterations in circulating tumor DNA and tumor-associated protein levels, which are commonly associated with cancer. It is performed on plasma derived from peripheral blood specimens.

SUMMARY:
This is a multi-site registry of patients receiving the Exact Sciences Multicancer Early Detection (MCED) test.

DETAILED DESCRIPTION:
This study was designed to simulate a real-world application of Exact Science's Multicancer Early Detection (MCED) test. Participants will be offered the Exact Science's MCED test annually for 3 years. If at any point during those 3 years a participant is diagnosed with cancer, they will become ineligible for further testing. Data will be collected for 5 years following the baseline test.

There will be two data collection approaches as part of this study. The first will be collection of self-report data related to the testing experience. The second will be periodic and largely automated extraction of pre-specified data elements from existing electronic data sources. A comparison data set will be constructed from records of individuals who did not receive the MCED test.

ELIGIBILITY:
Inclusion Criteria:

* Participant age at time of consent is between 50 and 80 years
* Agree to receive the Exact Sciences MCED test and follow-up imaging
* Willing and able to provide informed consent
* Access to a suitable technology and willing to complete surveys electronically

Exclusion Criteria:

* Any invasive tumor (excluding non-melanoma skin cancers) or hematological malignancy in the previous three years or current suspicion of cancer and/or in active treatment (e.g., chemotherapy, radiation therapy, immunotherapy, and/or surgery

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort will consist of particpants who have scheduled appointments with their primary health care provider at the participating clinics.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Vital status | Up to 5 years
  Particpant is alive or deceased
Cancer status | Up to 5 years
  Presence or absence of cancer

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz M Beer, MD, Principal Investigator — Exact Sciences
Locations (2):
- United States (2):
  - Endeavor Health, Evanston, Illinois
  - Baylor Scott & White Health, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study will be shared after de-identification. This may include text, tables, figures, and appendices. The study protocol, statistical analysis plan (when applicable), informed consent form (when applicable), and clinical study report (when applicable) will also be shared. Data will be shared with researchers who provide a methodologically sound proposal to achieve the aims outlined in the approved proposal.
Time Frame: Data will be available from 2 years and ending 4 years after publication.
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary Institutional Review Board (IRB)/Ethics Committee (EC) approvals or waivers as applicable to conduct research.